CLINICAL TRIAL: NCT00004266
Title: Randomized Study of Antihypertensives and Antilipemics in American Indians With Non-Insulin-Dependent Diabetes Mellitus at High Risk of Developing Nephropathy and Cardiovascular Disease
Brief Title: Drugs for High Blood Pressure and High Cholesterol in American Indians With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 199/11643; UMN-1967 (Other: Hennepin County Medical Center, Minneapolis); R01DK047112 (NIH)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Diabetic Nephropathy
Keywords: diabetic nephropathy; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Diabetic Nephropathies; Rare Diseases; Urogenital Diseases | interventions — Lisinopril; Nifedipine; Simvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nifedipine (Experimental): Daily nifedipine at a dose adjusted for high blood pressure. Cholestyramine or gemfibrozil is administered per National Cholesterol Education Program guidelines. Diuretics and doxazosin may be given concurrently.
  Interventions: Drug: Nifedipine
- Lisinopril (Experimental): Daily lisinopril at a dose adjusted for high blood pressure. Cholestyramine or gemfibrozil is administered per National Cholesterol Education Program guidelines. Diuretics and doxazosin may be given concurrently.
  Interventions: Drug: Lisinopril
- Nifedipine and simvastatin (Experimental): Daily nifedipine at a dose adjusted for high blood pressure, and simvastatin at a dose adjusted for high low-density lipoproteins. Supplemental cholestyramine may be given as needed. If cholestyramine is not tolerated or if triglycerides are high, gemfibrozil is substituted for cholestyramine.
  Interventions: Drug: Nifedipine; Drug: Simvastatin
- Lisinopril and simvastatin (Experimental): Lisinopril at a dose adjusted for high blood pressure and simvastatin at a dose adjusted for high low-density lipoproteins.
  Interventions: Drug: Lisinopril; Drug: Simvastatin

INTERVENTIONS:
Drug: Lisinopril
  Arms: Lisinopril; Lisinopril and simvastatin
Drug: Nifedipine
  Arms: Nifedipine; Nifedipine and simvastatin
Drug: Simvastatin
  Arms: Lisinopril and simvastatin; Nifedipine and simvastatin

SUMMARY:
OBJECTIVES:

I. Establish a long-term working relationship between clinical investigators and the Minnesota American Indian community.

II. Compare the effectiveness of lisinopril (an angiotensin-converting enzyme inhibitor) and nifedipine (a calcium channel blocker) in preventing nephropathy and vascular disease in Minnesota American Indians with non-insulin-dependent diabetes mellitus and microalbuminuria.

III. Compare the effectiveness of simvastatin (a 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor) with lipid-lowering strategies recommended by the National Cholesterol Education Program in preventing nephropathy and vascular diseases in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are randomly assigned to 1 of 4 treatment groups; therapy continues for 3 years. All patients receive instruction on diet, exercise, and smoking cessation.

The first group receives daily nifedipine at a dose adjusted for high blood pressure. Cholestyramine or gemfibrozil is administered per National Cholesterol Education Program guidelines. Diuretics and doxazosin may be given concurrently.

The second group receives daily lisinopril at a dose adjusted for high blood pressure. Cholestyramine or gemfibrozil is administered per National Cholesterol Education Program guidelines. Diuretics and doxazosin may be given concurrently.

The third group receives daily nifedipine at a dose adjusted for high blood pressure, and simvastatin at a dose adjusted for high low-density lipoproteins. Supplemental cholestyramine may be given as needed. If cholestyramine is not tolerated or if triglycerides are high, gemfibrozil is substituted for cholestyramine.

The fourth group receives lisinopril at a dose adjusted for high blood pressure and simvastatin at a dose adjusted for high low-density lipoproteins.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Non-insulin-dependent diabetes mellitus with documented fasting hyperglycemia Microalbuminuria OR clinically detectable albuminuria; Urine albumin excretion rate at least 30 mg/24 hours Low-density lipoproteins (fasting) at least 80 mg/dL Recruitment from American Indian population at Red Lake and Leech Lake reservations

--Prior/Concurrent Therapy-- At least 5 days since antihypertensives or antilipemics

--Patient Characteristics-- Renal: Urine albumin-to-creatinine ratio at least 30 mg/g; Creatinine clearance or estimated creatinine clearance at least 30 mL/min; No active urine sediment suggestive of glomerulonephritis, i.e.: No RBCs greater than 10/high-power field; No WBCs greater than 15/high-power field; No RBC casts

Cardiovascular: No symptomatic orthostatic hypotension; No poorly-compensated congestive heart failure; No requirement for angiotensin-converting enzyme inhibitors; No angina pectoris requiring nifedipine; No unstable angina; No episodes of angina occurring more than once a month; No chest pain of undetermined cause within 1 month; No severe hypertension requiring multiple antihypertensives; No myocardial infarction within 1 year; No stroke or transient ischemic attack within 1 year

Other: No known allergy to nifedipine, lisinopril, or simvastatin; No untreated proliferative retinopathy; Documented retinal exam within 1 year prior to entry; No alcohol or drug abuse affecting compliance; No other debilitating or acute illness; No pregnant or nursing women; Effective contraception required of fertile women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 1993-08 (Actual); Primary Completion 1999-07 (Actual); Study Completion 1999-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bertram L. Kasiske, Study Chair — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States